CLINICAL TRIAL: NCT01031706
Title: Sustained Impact of Hypertonic Saline on Mucociliary Clearance in Young Children With Cystic Fibrosis
Brief Title: Effect of Hypertonic Saline on Mucus Clearance in Children Ages 5-12 With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Scott Donaldson, MD, MD, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-1258; 1P50HL084934 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
Keywords: Hypertonic Saline; Pediatrics; Cystic Fibrosis; Mucociliary Clearance; Lung Clearance Index
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertonic saline (Experimental): 6% NaCl, 4 ml TID via eFlow
  Interventions: Drug: Hypertonic Saline
- Placebo (Placebo Comparator): 0.12% x 4ml via eFlow nebulizer
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hypertonic Saline — inhaled HS (6% NaCl, 4mL) three times a day for 28 days
  Other Names: HS
  Arms: Hypertonic saline
Drug: Placebo — 4 ml 0.12% NaCl inhaled three times a day x 28 days
  Other Names: .12% NaCl
  Arms: Placebo

SUMMARY:
Previous work demonstrated that inhaled hypertonic saline (HS) reduces exacerbation frequency and improves lung function in adults with cystic fibrosis (CF). It is unclear, however, whether HS will benefit young patients suffering from CF. The investigators propose to further support the concept that HS can benefit children with mild CF lung disease by performing a relatively short, placebo controlled study of HS in 5-12 year olds, using lung function and mucociliary clearance as key outcome measures.

DETAILED DESCRIPTION:
Our current understanding of the pathogenesis of CF lung disease stems from data that demonstrate the presence of airway surface liquid (ASL) dehydration in CF. ASL dehydration in CF is caused by defective chloride secretion through the cystic fibrosis transmembrane regulator (CFTR) and increased sodium reabsorption through the epithelial sodium channel (ENaC). ASL dehydration, in turn, interferes with the mucociliary clearance apparatus, causing a breach in a critical line of lung host defense. A number of novel therapeutics are now being developed to address this basic defect of disease, including the use of inhaled hypertonic saline.

Previous work demonstrated that inhaled hypertonic saline (HS) reduces exacerbation frequency and improves lung function in patients with clinically apparent lung disease. A number of issues revolving around the use of HS in CF remain unresolved. First, the typical patients enrolled in previous studies were adults (mean age = 26 yrs) with established lung disease (mean FEV1=78%). Despite our hypothesis that HS should positively affect MCC in preserved/normal airways, a common view of HS is that it benefits CF patients by inducing cough and transiently promoting the clearance of thick CF secretions. It has been questioned, therefore, whether HS will benefit patients who are younger and have mild (or undetectable) lung disease and potentially normal (though unmeasured) rates of MCC. Second, it is unclear whether the substantial beneficial effects of HS in CF were achieved because of a long (>4 hours) duration of action or in spite of an extremely short (~45 minutes) duration of action (the traditional view based upon experiments in normal epithelia). This issue is important, as it relates to the development and dosing of hydrator therapies that may have different pharmacodynamic profiles. Certainly, if twice daily dosing of a short acting compound is sufficient to provide significant clinical benefit, it would reduce the challenge of drug discovery for CF and ease the treatment burden imposed upon patients. The study of HS in CF provides us an opportunity to address this issue.

The hypothesis being tested is that HS will rehydrate CF airway secretions, producing a sustained acceleration in MCC in young children with CF, regardless of whether a measurable mucus clearance defect exists at this relatively early stage of disease. We predict a substantial acceleration of MCC will reduce the exacerbation rate in young children with CF. In addition, with the growing number of treatment modalities that are prescribed to patients with CF, adherence to complex and time consuming medical regimens becomes increasingly problematic and important. We therefore, wish to test an improved drug delivery platform for HS- the eFlow (Pari Pharma) vibrating mesh nebulizer, which has the potential to reduce treatment times, improve compliance, and increase treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Females or Males. If the subject is female and of childbearing potential (first menses has occurred), she must have a documented negative pregnancy test at screening and prior to each mucociliary clearance study. Those of childbearing potential must be abstinent or using an acceptable method of birth control (i.e. an Intrauterine Contraceptive Device with a failure rate of <1%, hormonal contraceptives or a barrier method).
* Age: 5-12 years, inclusive
* Diagnosis: Cystic fibrosis documented by a compatible clinical presentation and sweat chloride > 60 mEq/l or 2 disease causing CFTR mutations.
* Severity of the Disease: Suitable patients will have mild lung disease, as defined by:

  * Pulmonary Function: Each patient must have an FEV1 of greater than or equal to 60% of predicted at the screening visit.
  * Hemoglobin saturation: Patients must have an oxygen saturation of >92% on room air as determined by pulse oximetry at the screening visit.
* Informed consent - The patient and a parent or legally authorized guardian must agree to the subject's participation in the study by signing and dating the informed consent/assent forms after the nature of the study has been fully explained and all questions have been satisfactorily answered.

Exclusion Criteria:

* Unstable or asthmatic lung disease: As defined by a change in medical regimen during the preceding 2 weeks; an FEV1 15% below recent (within 6 months) clinical measurements. Patients with a history of co-existent asthma, as manifested by wheezing and significant bronchoreactivity (>15% increase in FEV1 with bronchodilator), will also be excluded.
* Other medication usage: Patients unable or unwilling to be withdrawn from hypertonic saline therapy for two weeks prior to Visit 1 (baseline MCC visit). Patients using Pulmozyme will be permitted to participate in this trial. Patients on chronic, cycling antibiotics will be required to have completed at least 2 full cycles of the prescribed antibiotic prior to enrollment and should not cycle on or off this therapy during the treatment period of the study.
* Spirometry Performance: Those subjects who are unable to perform acceptable, reproducible spirometry will be excluded from this study.
* Drug allergy: A history of allergy or intolerance to any of the study medications, including albuterol or hypertonic saline.
* Have received an investigational drug or therapy during the preceding 30 days.
* Have had radiation exposure within the past year that would cause them to exceed Federal Regulations by participating in this study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elkins MR, Robinson M, Rose BR, Harbour C, Moriarty CP, Marks GB, Belousova EG, Xuan W, Bye PT; National Hypertonic Saline in Cystic Fibrosis (NHSCF) Study Group. A controlled trial of long-term inhaled hypertonic saline in patients with cystic fibrosis. N Engl J Med. 2006 Jan 19;354(3):229-40. doi: 10.1056/NEJMoa043900. PMID 16421364
- [Background] Donaldson SH, Bennett WD, Zeman KL, Knowles MR, Tarran R, Boucher RC. Mucus clearance and lung function in cystic fibrosis with hypertonic saline. N Engl J Med. 2006 Jan 19;354(3):241-50. doi: 10.1056/NEJMoa043891. PMID 16421365
- [Background] Bennett WD, Olivier KN, Zeman KL, Hohneker KW, Boucher RC, Knowles MR. Effect of uridine 5'-triphosphate plus amiloride on mucociliary clearance in adult cystic fibrosis. Am J Respir Crit Care Med. 1996 Jun;153(6 Pt 1):1796-801. doi: 10.1164/ajrccm.153.6.8665037.
- [Background] Matsui H, Grubb BR, Tarran R, Randell SH, Gatzy JT, Davis CW, Boucher RC. Evidence for periciliary liquid layer depletion, not abnormal ion composition, in the pathogenesis of cystic fibrosis airways disease. Cell. 1998 Dec 23;95(7):1005-15. doi: 10.1016/s0092-8674(00)81724-9. PMID 9875854
- [Background] Tarran R. Regulation of airway surface liquid volume and mucus transport by active ion transport. Proc Am Thorac Soc. 2004;1(1):42-6. doi: 10.1513/pats.2306014. PMID 16113411
- [Background] Elkins MR, Bye PT. Inhaled hypertonic saline as a therapy for cystic fibrosis. Curr Opin Pulm Med. 2006 Nov;12(6):445-52. doi: 10.1097/01.mcp.0000245714.89632.b2. PMID 17053496
- [Background] Modi AC, Quittner AL. Validation of a disease-specific measure of health-related quality of life for children with cystic fibrosis. J Pediatr Psychol. 2003 Dec;28(8):535-45. doi: 10.1093/jpepsy/jsg044. PMID 14602844
- [Derived] Donaldson SH, Danielle Samulski T, LaFave C, Zeman K, Wu J, Trimble A, Ceppe A, Bennett WD, Davis SD. A four week trial of hypertonic saline in children with mild cystic fibrosis lung disease: Effect on mucociliary clearance and clinical outcomes. J Cyst Fibros. 2020 Nov;19(6):942-948. doi: 10.1016/j.jcf.2020.07.009. Epub 2020 Jul 12. PMID 32669217

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypertonic Saline | Placebo
Started | 14 | 9
Completed | 12 | 8
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Number of subjects passing screening
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline | Placebo | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (3.3) | 9.8 (3.6) | 11.1 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Mucociliary Clearance Rate
Description: Average radio tracer clearance through 90 minutes (MCC90) is primary index of mucociliary clearance at each study.
  Primary study outcome: is absolute change in MCC90 between baseline and at end of treatment (where MCC measured 8-12 hours after final dose of study drug) - reflects sustained impact on MCC
Time Frame: Baseline versus after completion of 4 week treatment period
Population: All subjects with available data analyzed
Measure: Mean (Standard Error); unit: percent clearance
Arm/Group | Hypertonic Saline | Placebo
Number analyzed (Participants) | 12 | 8
percent clearance | 2.77 (.98) | -2.35 (1.82)

2. Secondary Outcome: FEV1 (Spirometry) Change
Description: Absolute change in % predicted FEV1 between baseline and after 4 weeks of treatment calculated
Time Frame: Baseline and after 4 weeks of treatment
Population: All available data included. Carry-forward of last FEV1 value (after 2 weeks of treatment) performed when data at 4 week time point not available
Measure: Mean (Standard Error); unit: Percentage of predicted FEV1
Arm/Group | Hypertonic Saline | Placebo
Number analyzed (Participants) | 13 | 8
Percentage of predicted FEV1 | 3.38 (2.01) | 1.09 (3.19)

ADVERSE EVENTS:
Time Frame: 1 month
Description: All events between screening and end of treatment recorded. At start of each visit, subject is asked whether they have experienced any new symptoms or problems since the prior visit.
Arm/Group | Hypertonic Saline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 11/14 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypertonic Saline (N=14) | Placebo (N=9)
Cough during study drug inhalation (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Increased Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 6 (7)
Increased sputum production (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cystic Fibrosis exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
New Pulmonary Pathogen (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) — Re-aquisition of pseudmonas after prolonged negative culture; new Mycobacterium abscessus on culture
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1)
worsened steatorhea (Gastrointestinal disorders) | 2 (3) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
fever (General disorders) | 1 (1) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (3)
headache (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Hyperactivity (General disorders) | 0 (0) | 1 (1)
Pharynx irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Otalgia (Ear and labyrinth disorders) | 1 (1) | 0 (0)
nasal/sinus congestions (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes